CLINICAL TRIAL: NCT06754592
Title: Role of Dynamic Ultrasound in Assessment of Shoulder Impingement Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Robier Isaac Ibrahim, Role of dynamic Ultrasound in assessment of shoulder impingement syndrome, Sohag University
Other Study IDs: Soh-Med--24-12-11MS
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound — evaluate the effectiveness of dynamic high-resolution ultrasonography in identifying various abnormalities of the shoulder impingement syndrome, especially the subacromial type, and to determine the added value of dynamic ultrasonography compared to static examination of such cases. Furthermore, we will compare these findings to MRI
  Other Names: MRI

SUMMARY:
This study aims to evaluate the effectiveness of dynamic high-resolution ultrasonography in identifying various abnormalities of the shoulder impingement syndrome, especially the subacromial type, and to determine the added value of dynamic ultrasonography compared to static examination of such cases. Furthermore, we will compare these findings to MRI, which we regard as the standard in our cases.

DETAILED DESCRIPTION:
Patients with shoulder impingement syndrome often experience pain primarily in the anterior and lateral areas of the acromion, which can radiate to the lateral aspect of the mid-arm. This pain typically worsens at night and when lying on the affected side. Additionally, some patients may experience stiffness and weakness due to the pain.

When assessing a patient with signs of impingement, it is essential to evaluate the condition of the rotator cuff and the extent of any tears. This information allows surgeons to create an effective strategy for ongoing patient management.

Ultrasound (US) and magnetic resonance imaging (MRI) are effective tools for diagnosing rotator cuff disorders, especially when it comes to detecting full-thickness rotator cuff tears, due to their high sensitivity. However, their overall sensitivity for identifying partial rotator cuff tears and tendinopathy is lower. Impingement-related conditions, such as bursitis and changes or ruptures in tendons, can be visualized using a linear sonography.

Ultrasound (US) offers several advantages over MRI. One key benefit is that ultrasonography is a dynamic form of imaging, while MRI provides static images. US is also portable, better tolerated by patients, and allows for direct interaction with patients; this enables patients to point to the symptomatic area, which can enhance diagnostic accuracy. Additionally, ultrasound is less time-consuming, more cost-effective, and more readily available in secondary and tertiary care settings compared to MRI.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients present with shoulder pain with positive clinical tests suggestive of shoulder impingement syndrome

Exclusion Criteria:

* History of shoulder surgery, instability disorders, shoulder girdle fracture, radiation therapy to the shoulder, neoplastic lesions, and congenital anomalies of the shoulder. Patients having contraindications to perform MRI (Patients with electrically, magnetically, or mechanically activated implants, pacemakers, cochlear implants, or any metallic orthopedic implants) and claustrophobic patients).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: male and female patients present with shoulder pain with positive clinical tests suggestive of shoulder impingement syndrome
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12-26 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison between Ultrasound findings and Magnetic Resonance Imaging findings in patients with clinical diagnosis of Shoulder Impingement Syndrome | Baseline
  Evaluate the effectiveness of dynamic high-resolution ultrasonography in identifying various abnormalities of the shoulder impingement syndrome and to compare these findings to MRI, which we regard as the standard in our cases

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided